CLINICAL TRIAL: NCT01340027
Title: A Randomized, Double-Blind, Factorial, Parallel-Group, Active and Placebo-Controlled, Multicenter Dose-Ranging Study to Evaluate the Efficacy, Safety and Tolerability of Six Dose Combinations of Solifenacin Succinate and Mirabegron Compared to Mirabegron and Solifenacin Succinate Monotherapies in the Treatment of Overactive Bladder.
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of Mirabegron and Solifenacin Succinate Alone and in Combination for the Treatment of Overactive Bladder
Acronym: Symphony
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 178-CL-100; 2010-020601-32 (EudraCT Number)
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urologic Diseases; Urinary Bladder Diseases; Urological Manifestations; Signs and Symptoms; Urinary Bladder, Overactive
Keywords: Urinary incontinence; Overactive bladder (OAB); Micturition; Frequency; YM178; Urgency incontinence; Urgency
MeSH Terms: conditions — Urologic Diseases; Urinary Bladder Diseases; Urological Manifestations; Signs and Symptoms; Urinary Bladder, Overactive; Urinary Incontinence | interventions — mirabegron; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Placebo (Placebo Comparator): Participants received matching placebo tablets orally once a day for 12 weeks
  Interventions: Drug: Placebo
- Mirabegron 25 mg (Active Comparator): Participants received mirabegron 25 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Mirabegron
- Mirabegron 50 mg (Active Comparator): Participants received mirabegron 50 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Mirabegron
- Solifenacin 2.5 mg (Active Comparator): Participants received solifenacin 2.5 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Solifenacin succinate
- Solifenacin 5 mg (Active Comparator): Participants received solifenacin 5 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Solifenacin succinate
- Solifenacin 10 mg (Active Comparator): Participants received solifenacin 10 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Solifenacin succinate
- Solifenacin 2.5 mg and Mirabegron 25 mg (Experimental): Participants received solifenacin 2.5 mg and mirabegron 25 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Mirabegron; Drug: Solifenacin succinate
- Solifenacin 2.5 mg and Mirabegron 50 mg (Experimental): Participants received solifenacin 2.5 mg and mirabegron 50 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Mirabegron; Drug: Solifenacin succinate
- Solifenacin 5 mg and Mirabegron 25 mg (Experimental): Participants received solifenacin 5 mg and mirabegron 25 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Mirabegron; Drug: Solifenacin succinate
- Solifenacin 5 mg and Mirabegron 50 mg (Experimental): Participants received solifenacin 5 mg and mirabegron 50 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Mirabegron; Drug: Solifenacin succinate
- Solifenacin 10 mg and Mirabegron 25 mg (Experimental): Participants received solifenacin 10 mg and mirabegron 25 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Mirabegron; Drug: Solifenacin succinate
- Solifenacin 10 mg and Mirabegron 50 mg (Experimental): Participants received solifenacin 10 mg and mirabegron 50 mg tablets orally once a day for 12 weeks
  Interventions: Drug: Mirabegron; Drug: Solifenacin succinate

INTERVENTIONS:
Drug: Mirabegron — oral
  Other Names: Betmiga; Myrbetric; Myrbetriq; Betanis; YM178
  Arms: Mirabegron 25 mg; Mirabegron 50 mg; Solifenacin 10 mg and Mirabegron 25 mg; Solifenacin 10 mg and Mirabegron 50 mg; Solifenacin 2.5 mg and Mirabegron 25 mg; Solifenacin 2.5 mg and Mirabegron 50 mg; Solifenacin 5 mg and Mirabegron 25 mg; Solifenacin 5 mg and Mirabegron 50 mg
Drug: Solifenacin succinate — oral
  Other Names: Vesikur; Vesicare
  Arms: Solifenacin 10 mg; Solifenacin 10 mg and Mirabegron 25 mg; Solifenacin 10 mg and Mirabegron 50 mg; Solifenacin 2.5 mg; Solifenacin 2.5 mg and Mirabegron 25 mg; Solifenacin 2.5 mg and Mirabegron 50 mg; Solifenacin 5 mg; Solifenacin 5 mg and Mirabegron 25 mg; Solifenacin 5 mg and Mirabegron 50 mg
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine how well two medicines in combination (solifenacin succinate and mirabegron) work in the treatment of bladder problems over a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria at Visit 1/Screening:

  * Subject has a Body Mass Index (BMI) of between 18 and 35 kg/m^2 and a total body weight between 50 and 95 kg;
  * Subject is willing and able to complete the micturition diary and questionnaires correctly and is willing and able to measure his/her vital signs at home at stipulated time points, using the device provided by the study personnel, and to adequately record the readings;
  * Subject has symptoms of overactive bladder (OAB; urinary frequency, urgency and/or urgency incontinence) for at least 3 months.
* Inclusion Criteria at Visit 3/Baseline:

  * Subject has experienced frequency of micturition on average ≥ 8 times per 24-hour period during the 3-day micturition diary period (incontinence episode should not be counted as a micturition);
  * Subject must experience at least 1 episode of urgency (grade 3 or 4) per 24-hour period (with or without urgency incontinence) during the 3 day micturition diary period.

Exclusion Criteria:

* Exclusion Criteria at Visit 1/Screening:

  * Subject is breastfeeding, pregnant or intends to become pregnant during the study. The pregnancy test (Beta Human Chorionic Gonadotropin in serum) at Screening must be negative in women of childbearing potential;
  * Female subjects of childbearing potential and not using a highly effective method of birth control during the study and for 30 days after final study drug administration.
  * Male subjects (unless surgically sterile) with female spouses/partners who are of childbearing potential, and not using a barrier method of contraception during the study and for 30 days after final study drug administration. In addition, female spouses/partners of male subjects and who are of childbearing potential should also use a highly effective method of birth control during the study and for 30 days after final study drug administration. Highly effective methods of birth control are defined as those, alone or in combination, that result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly.
  * Subject has significant post-void residual (PVR) volume (> 150 mL);
  * Subject has significant stress incontinence or mixed stress/urgency incontinence where stress is the predominant factor as determined by the Investigator (for female subjects confirmed by the cough provocation test);
  * Subject has a neurological cause for detrusor overactivity;
  * Subject has an indwelling catheter or practices intermittent self-catheterization;
  * Subject has diabetic neuropathy;
  * Subject has chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs;
  * Subject has had previous lower urinary tract or pelvic floor surgery (except cystoscopy);
  * Subject has had intravesical treatment in the past 12 months with e.g., botulinum toxin, resiniferatoxin, capsaicin;
  * Subject has uncontrolled narrow angle glaucoma, urinary or gastric retention, severe ulcerative colitis or Crohn's Disease, toxic megacolon, myasthenia gravis or any other condition which makes the use of anticholinergics contraindicated;
  * Subject has clinically significant cardiovascular or cerebrovascular diseases within 6 months prior to Screening, such as myocardial infarction, uncontrolled angina, significant ventricular arrhythmias, heart failure and stroke;
  * Subject is receiving current non-drug treatment including electro-stimulation therapy (with the exception of a bladder training program or pelvic floor exercises which started more than 30 days prior to Screening);
  * Subject is using medications intended to treat OAB or prohibited medications.
  * Subject has known or suspected hypersensitivity to solifenacin succinate, mirabegron or any of their excipients;
  * Subject has any significant neurological disease or defect affecting bladder function (e.g., neurogenic bladder, systemic or central neurological disease such as multiple sclerosis [MS] and Parkinson's disease);
  * Subject has severe hypertension which is defined as a sitting average systolic blood pressure ≥ 180 mmHg and/or an average diastolic blood pressure ≥ 110 mmHg;
* Exclusion Criteria at Visit 2/Placebo Run-In:

  * Subject has evidence of a urinary tract infection (UTI) (urine culture containing > 100,000 cfu/mL). The subject can be enrolled into the study after successful treatment of the UTI (confirmed by a laboratory result of negative urine culture). However, the subject must be re screened if the initial screening visit was > 28 days;
  * Subject has a QT interval > 450 ms or is at risk of QT prolongation (e.g., family history of long QT syndrome, hypokalaemia) or is on drug treatment known to be associated with QT prolongation;
  * Subject has clinically significant abnormalities on the 12 lead electrocardiogram (ECG);
  * Subject has serum creatinine > 150 µmol/L, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2x upper limit of normal (ULN), gamma-glutamyltransferase (γ-GT) > 3x ULN, or total bilirubin > 2x ULN, as assessed in Screening samples;
* Exclusion Criteria at Visit 3/Baseline:

  * Subject had an average total daily urine volume > 3000 mL as recorded in the micturition diary period;
  * Subject has severe hypertension which is defined as a sitting average systolic blood pressure ≥ 180 mmHg and/or an average diastolic blood pressure ≥ 110 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1307 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2012-06-28 (Actual); Study Completion 2012-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Astellas Pharma Europe B.V.; Principal Investigator, Principal Investigator — Bristol Urological Institute
Locations (133):
- Belarus (4):
  - BY37101, Minsk
  - BY37102, Minsk
  - BY37103, Minsk
  - BY37104, Vitebsk
- Belgium (4):
  - BE32102, Brussels
  - BE32104, Edegem
  - BE32103, Ghent
  - BE32101, Leuven
- Czechia (10):
  - CZ42005, Bohumín
  - CZ42003, Hradec Králové
  - CZ42011, Ostrava
  - CZ42006, Pilsen
  - CZ42001, Prague
  - CZ42007, Prague
  - CZ42009, Prague
  - CZ42010, Roudnice nad Labem
  - CZ42012, Sternberk
  - CZ42002, Uherské Hradiště
- Denmark (3):
  - DK45101, Aarhus N
  - DK45102, Herlev
  - DK45104, Holstebro
- Finland (4):
  - FI35803, Helsinki
  - FI35804, Kouvola
  - FI35801, Oulu
  - FI35802, Tampere
- France (7):
  - FR33104, Colmar
  - FR33108, Dijon
  - FR33103, Orléans
  - FR33111, Paris
  - FR33112, Paris
  - FR33106, Toulouse
  - FR33110, Tours
- Germany (10):
  - DE49109, Bad Ems
  - DE49103, Göttingen
  - DE49117, Hagenow
  - DE49105, Hettstedt
  - DE49108, Leipzig
  - DE49110, Neustadt in Sachsen
  - DE49118, Reutlingen
  - DE49101, Rostock
  - DE49111, Sangerhausen
  - DE49104, Wismar
- Hungary (7):
  - HU36108, Csongrád
  - HU36101, Győr
  - HU36106, Körmend
  - HU36110, Miskolc
  - HU36104, Sopron
  - HU36103, Szekszárd
  - HU36107, Tatabánya
- Italy (4):
  - IT39103, Avellino
  - IT39101, Catanzaro
  - IT39105, Florence
  - IT39102, Treviglio (BG)
- Netherlands (4):
  - NL31104, Amsterdam
  - NL31106, Maastricht
  - NL31102, Sneek
  - NL31101, Winterswijk
- Norway (2):
  - NO47104, Elverum
  - NO47102, Hamar
- Poland (9):
  - PL48107, Krakow
  - PL48103, Lodz
  - PL48108, Lublin
  - PL48106, Piaseczno
  - PL48104, Puławy
  - PL48101, Warsaw
  - PL48105, Warsaw
  - PL48112, Więcbork
  - PL48111, Wroclaw
- Portugal (7):
  - PT35102, Coimbra
  - PT35105, Coimbra
  - PT35104, Lisbon
  - PT35107, Lisbon
  - PT35110, Porto
  - PT35101, Porto
  - PT35106, Tomar
- Romania (8):
  - RO40106, Brasov
  - RO40102, Bucharest
  - RO40104, Bucharest
  - RO40103, Bucharest
  - RO40108, Bucharest
  - RO40101, Craiova
  - RO40105, Craiova
  - RO40107, Sibiu
- Russia (10):
  - RU70112, Kazan'
  - RU70108, Moscow
  - RU70110, Moscow
  - RU70102, Saint Petersburg
  - RU70103, Saint Petersburg
  - RU70106, Saint Petersburg
  - RU70101, Saint Petersburg
  - RU70107, Saint Petersburg
  - RU70109, Saint Petersburg
  - RU70113, Ufa
- Slovakia (11):
  - SK42109, Banská Bystrica
  - SK42112, Bratislava
  - SK42107, Košice
  - SK42113, Malacky
  - SK42104, Nitra
  - SK42105, Pieštany
  - SK42106, Piešťany
  - SK42102, Prešov
  - SK42108, Trenčín
  - SK42101, Trenčín
  - SK42103, Žilina
- Spain (7):
  - ES34103, Madrid
  - ES34101, Madrid
  - ES34109, Madrid
  - ES34102, Madrid
  - ES34105, Pamplona
  - ES34104, Sant Joan d'Alacant
  - ES34107, Seville
- Sweden (5):
  - SE46101, Gothenburg
  - SE46103, Karlshamn
  - SE46104, Malmo
  - SE46102, Stockholm
  - SE46105, Tanumshede
- Ukraine (8):
  - UA38104, Dnipro
  - UA38102, Donetsk
  - UA38111, Donetsk
  - UA38106, Kiev
  - UA38109, Kiev
  - UA38107, Lviv
  - UA38101, Odesa
  - UA38103, Zaporizhzhya
- United Kingdom (9):
  - GB44103, Bristol
  - GB44108, Cambridge
  - GB44106, Garston
  - GB44111, Glasgow
  - GB44104, Nantwich
  - GB44110, Northwood
  - GB44107, Plymouth
  - GB44101, Reading
  - GB44105, Sandbach

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Abrams P, Kelleher C, Staskin D, Rechberger T, Kay R, Martina R, Newgreen D, Paireddy A, van Maanen R, Ridder A. Combination treatment with mirabegron and solifenacin in patients with overactive bladder: efficacy and safety results from a randomised, double-blind, dose-ranging, phase 2 study (Symphony). Eur Urol. 2015 Mar;67(3):577-88. doi: 10.1016/j.eururo.2014.02.012. Epub 2014 Feb 19. PMID 24612659
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female patients with symptoms of overactive bladder (OAB; urgency, urinary frequency and/or urgency incontinence) for at least 3 months. The study was conducted at 141 sites in 20 countries in Europe.
Pre-assignment Details: After screening, 1658 participants entered a 2-week, single-blind, placebo run-in period. After completion of the run-in period, 1307 participants were randomly assigned to 1 of the 12 treatment arms in a 1:1:1:1:2:1:2:2:2:2:1:1 ratio.
Groups:
- Solifenacin 2.5 mg + Mirabegron 25 mg: Participants received solifenacin 2.5 mg and mirabegron 25 mg tablets orally once a day for 12 weeks.
- Solifenacin 2.5 mg + Mirabegron 50 mg: Participants received solifenacin 2.5 mg and mirabegron 50 mg tablets orally once a day for 12 weeks.
- Solifenacin 5 mg + Mirabegron 25 mg: Participants received solifenacin 5 mg and mirabegron 25 mg tablets orally once a day for 12 weeks.
- Solifenacin 5 mg + Mirabegron 50 mg: Participants received solifenacin 5 mg and mirabegron 50 mg tablets orally once a day for 12 weeks.
- Solifenacin 10 mg + Mirabegron 25 mg: Participants received solifenacin 10 mg and mirabegron 25 mg tablets orally once a day for 12 weeks.
- Solifenacin 10 mg + Mirabegron 50 mg: Participants received solifenacin 10 mg and mirabegron 50 mg tablets orally once a day for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Started | 81 | 78 | 79 | 79 | 156 | 78 | 149 | 149 | 144 | 152 | 81 | 81
Received Treatment | 81 | 78 | 78 | 79 | 156 | 78 | 149 | 149 | 144 | 152 | 81 | 81
Completed | 76 | 71 | 75 | 75 | 146 | 74 | 142 | 142 | 136 | 146 | 79 | 77
Not Completed | 5 | 7 | 4 | 4 | 10 | 4 | 7 | 7 | 8 | 6 | 2 | 4
Not completed — Randomized but Never Received Study Drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 1 | 2 | 2 | 1 | 4 | 1 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0 | 6 | 0 | 0 | 1 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 1 | 3 | 3 | 2 | 3 | 4 | 1 | 2 | 0 | 1
Not completed — Miscellaneous | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Measure data are provided for all randomized patients who took at least 1 dose of double-blind study drug (Safety Analysis Set). One participant randomized to the Mirabegron 25 mg arm received treatment with Solifenacin 5 mg + Mirabegron 50 mg in error and is counted in that arm for safety analysis set analyses.
Groups:
- Solifenacin 2.5 mg +Mirabegron 25 mg: Participants received solifenacin 2.5 mg and mirabegron 25 mg tablets orally once a day for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg +Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg | Total
Number analyzed (Participants) | 81 | 77 | 78 | 79 | 156 | 78 | 149 | 149 | 144 | 153 | 81 | 81 | 1306
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (13.37) | 55.2 (14.45) | 53.4 (13.98) | 56.1 (11.71) | 54.2 (15.53) | 55.0 (12.82) | 55.8 (13.82) | 53.7 (14.55) | 55.0 (14.57) | 54.1 (14.09) | 56.5 (12.34) | 55.5 (13.82) | 54.8 (13.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 52 | 52 | 51 | 103 | 53 | 100 | 100 | 95 | 101 | 52 | 54 | 867
  Male | 27 | 25 | 26 | 28 | 53 | 25 | 49 | 49 | 49 | 52 | 29 | 27 | 439
Race/Ethnicity, Customized [Number; unit: participants]
  White | 81 | 77 | 78 | 78 | 156 | 77 | 149 | 148 | 143 | 153 | 81 | 81 | 1302
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type of Overactive Bladder (OAB) [Number; unit: participants]
  Urge Incontinence | 14 | 27 | 19 | 18 | 39 | 19 | 42 | 33 | 35 | 35 | 23 | 20 | 324
  Mixed | 9 | 10 | 10 | 10 | 27 | 11 | 22 | 20 | 19 | 18 | 14 | 10 | 180
  Frequency | 56 | 39 | 48 | 50 | 89 | 48 | 84 | 95 | 90 | 100 | 44 | 50 | 793
  Missing | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 9
Duration of OAB Symptoms [Mean (Standard Deviation); unit: months] | 48.3 (38.37) | 61.2 (68.03) | 56.9 (66.62) | 60.2 (67.85) | 61.8 (78.21) | 52.4 (56.98) | 57.7 (68.91) | 57.0 (66.85) | 56.3 (84.78) | 57.4 (81.53) | 64.9 (100.57) | 57.4 (80.12) | 57.8 (73.82)
Mean Number of Micturitions per 24 Hours [Mean (Standard Deviation); unit: micturitions] — The average number of micturitions (urinations) a day recorded by the participant in a micturition diary for 3 days prior to the Baseline visit. Data available for 81, 76, 78, 79, 155, 78, 149, 148, 144, 152, 81 and 81 participants in each treatment arm respectively.
  micturitions | 10.36 (2.036) | 11.29 (2.581) | 10.78 (2.254) | 11.10 (3.056) | 11.34 (3.158) | 11.29 (2.896) | 11.25 (3.643) | 11.00 (2.260) | 10.92 (2.386) | 11.25 (3.171) | 11.14 (2.268) | 11.24 (2.453) | 11.10 (2.794)
Mean Volume Voided per Micturition [Mean (Standard Deviation); unit: mL] — Recorded by the patient in a micturition diary for 3 days prior to the Baseline visit. Data available for 81, 76, 78, 79, 155, 78, 149, 148, 144, 152, 81 and 81 participants in each treatment arm respectively.
  mL | 156.4 (52.80) | 152.7 (56.70) | 156.8 (52.33) | 162.4 (57.59) | 145.5 (59.34) | 148.0 (52.74) | 156.8 (61.97) | 149.8 (50.05) | 155.0 (55.55) | 153.1 (51.88) | 141.4 (51.29) | 155.3 (62.13) | 152.5 (55.65)
Mean Number of Urgency Episodes per 24 Hours [Mean (Standard Deviation); unit: urgency episodes] — Urgency episodes were those classified by the participant in a 3-day micturition diary as 3 or 4 on the Patient Perception of Intensity of Urgency (PPIUS) scale: 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet. Data available for 81, 76, 78, 79, 155, 78, 149, 148, 144, 152, 81 and 81 participants in each treatment arm respectively.
  urgency episodes | 5.26 (3.079) | 6.25 (3.332) | 6.58 (3.981) | 6.20 (3.870) | 6.41 (4.154) | 6.37 (4.530) | 6.05 (3.749) | 6.78 (3.419) | 6.26 (3.928) | 6.49 (4.238) | 6.91 (4.319) | 6.81 (4.312) | 6.37 (3.931)
Mean Level of Urgency [Mean (Standard Deviation); unit: units on a scale] — Average of participants' ratings on the degree of associated urgency for each micturition and/or incontinence episode recorded in a 3-day micturition diary according to the following 5-point categorical scale (Patient Perception of Intensity of Urgency Scale): 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet. Data available for 81, 76, 78, 79, 155, 78, 149, 148, 144, 152, 81 and 81 participants in each treatment arm respectively.
  units on a scale | 2.45 (0.503) | 2.53 (0.439) | 2.55 (0.508) | 2.53 (0.539) | 2.49 (0.508) | 2.48 (0.503) | 2.49 (0.445) | 2.59 (0.446) | 2.50 (0.491) | 2.51 (0.441) | 2.57 (0.493) | 2.53 (0.473) | 2.52 (0.479)
Mean Number of Nocturia Episodes per 24 Hours [Mean (Standard Deviation); unit: nocturia episodes] — The average number of times a participant woke at night to urinate (excluding incontinence only episodes) recorded for 3 days prior to the Baseline visit in the patient micturition diary. Data available for 81, 76, 78, 79, 155, 78, 149, 148, 144, 152, 81 and 81 participants in each treatment arm respectively.
  nocturia episodes | 2.19 (1.584) | 2.18 (1.392) | 2.31 (1.517) | 2.46 (1.852) | 2.19 (1.399) | 2.50 (1.859) | 2.64 (2.259) | 2.05 (1.219) | 2.28 (1.449) | 2.27 (1.305) | 2.65 (2.525) | 2.41 (2.001) | 2.33 (1.701)
Mean Number of Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: incontinence episodes] — The average number of incontinence episodes (any involuntary leakage of urine) a day recorded by the participant in a micturition diary for 3 days prior to the Baseline visit. Data are reported for participants who took at least 1 dose of double-blind study medication with available primary efficacy data who reported at least 1 incontinence episode in the Baseline diary (Full Analysis Set-Incontinence): 17, 13, 18, 15, 35, 15, 35, 33, 32, 24, 24, 20 participants in each treatment arm respectively.
  incontinence episodes | 0.95 (0.765) | 1.87 (1.578) | 1.26 (1.000) | 1.80 (1.167) | 1.33 (1.242) | 1.40 (1.280) | 1.27 (1.096) | 1.14 (0.791) | 1.24 (1.108) | 1.17 (1.196) | 1.53 (1.235) | 1.25 (0.858) | 1.31 (1.109)
Mean Number of Urgency Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: urgency incontinence episodes] — The average number of urgency incontinence episodes (involuntary urine leakage accompanied by or immediately preceded by urgency) a day recorded by the participant in a micturition diary for 3 days prior to the Baseline visit. Data are reported for participants who took at least 1 dose of double-blind study medication with available primary efficacy data who reported at least 1 incontinence episode in the Baseline diary (Full Analysis Set-Incontinence): 17, 13, 18, 15, 35, 15, 35, 33, 32, 24, 24, and 20 participants in each treatment arm respectively.
  urgency incontinence episodes | 0.78 (0.807) | 1.54 (1.337) | 1.19 (1.043) | 1.56 (1.052) | 1.32 (1.227) | 1.18 (1.308) | 0.96 (0.903) | 1.06 (0.757) | 1.23 (1.118) | 1.08 (1.193) | 1.51 (1.247) | 1.20 (0.901) | 1.20 (1.072)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (EOT) in Mean Volume Voided Per Micturition
Description: The average volume voided per micturition was calculated from the volume of each micturition measured by the participant and recorded in a micturition diary for 3 days before the Baseline and Week 12 clinic visits.
Time Frame: Baseline and Week 12
Population: The Full Analysis Set (FAS) comprised all participants took at least 1 dose of double-blind study medication after randomization and had primary efficacy data (mean volume voided) derived from the diary at Baseline and at least 1 post-baseline visit. Last observation carried forward imputation (LOCF) was utilized.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
mL | 14.0 (5.91) | 24.9 (6.06) | 34.5 (6.02) | 36.4 (6.02) | 36.0 (4.32) | 36.2 (6.06) | 39.4 (4.37) | 41.9 (4.36) | 53.6 (4.45) | 54.2 (4.31) | 57.6 (5.99) | 62.3 (5.90)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; Statistical comparisons were made using 2-sided tests at the 0.05 significance level. No adjustment for multiple testing was performed. The ANCOVA model for all pairwise comparisons includes the 2 main factors mirabegron dose and solifenacin succinate dose and their interaction, sex, age group and geographic region as fixed factors and Baseline value as a covariate. Least squares (LS) mean differences were calculated by subtracting Solifenacin 5 mg/Placebo from the comparison treatment group; Test type: Superiority or Other; p = 0.97, ANCOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-14.3 to 14.9], Standard Error of Mean 7.44
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.58, ANCOVA; LS Mean Difference = 3.4, 95% CI 2-sided [-8.6 to 15.5], Standard Error of Mean 6.15
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.33, ANCOVA; LS Mean Difference = 5.9, 95% CI 2-sided [-6.1 to 18.0], Standard Error of Mean 6.13
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = 17.6, 95% CI 2-sided [5.4 to 29.8], Standard Error of Mean 6.20
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = 18.2, 95% CI 2-sided [6.2 to 30.2], Standard Error of Mean 6.10
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = 21.7, 95% CI 2-sided [7.2 to 36.1], Standard Error of Mean 7.37
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 26.3, 95% CI 2-sided [11.9 to 40.7], Standard Error of Mean 7.32
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.20, ANCOVA; LS Mean Difference = 11.0, 95% CI 2-sided [-5.6 to 27.6], Standard Error of Mean 8.46
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.015, ANCOVA; LS Mean Difference = 20.5, 95% CI 2-sided [4.0 to 37.1], Standard Error of Mean 8.43
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = 22.4, 95% CI 2-sided [5.9 to 39.0], Standard Error of Mean 8.43
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = 22.0, 95% CI 2-sided [7.6 to 36.3], Standard Error of Mean 7.32
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.009, ANCOVA; LS Mean Difference = 22.2, 95% CI 2-sided [5.6 to 38.8], Standard Error of Mean 8.46
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 25.4, 95% CI 2-sided [11.0 to 39.8], Standard Error of Mean 7.35
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 27.9, 95% CI 2-sided [13.5 to 42.3], Standard Error of Mean 7.34
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 39.6, 95% CI 2-sided [25.1 to 54.1], Standard Error of Mean 7.39
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean DIfference = 40.2, 95% CI 2-sided [25.8 to 54.5], Standard Error of Mean 7.31
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 43.6, 95% CI 2-sided [27.1 to 60.1], Standard Error of Mean 8.42
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 48.3, 95% CI 2-sided [31.9 to 64.7], Standard Error of Mean 8.35

2. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Micturitions Per 24 Hours
Description: The average number of micturitions (urinations) per 24 hours was derived from the number of urinations (excluding incontinence only episodes) per day recorded by the participant in the micturition diary for 3-days before the Baseline and Week 12 clinic visits.
Time Frame: Baseline and Week 12
Population: Full analysis set; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
micturitions | -2.43 (0.291) | -2.48 (0.298) | -2.56 (0.296) | -2.44 (0.296) | -2.54 (0.212) | -3.22 (0.298) | -2.58 (0.215) | -2.93 (0.215) | -2.56 (0.219) | -3.34 (0.212) | -3.42 (0.294) | -3.52 (0.291)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; Statistical comparisons were made using 2-sided tests at the 0.05 significance level. No adjustment for multiple testing was performed. The ANCOVA model for all pairwise comparisons includes the 2 main factors mirabegron dose and solifenacin succinate dose and their interaction, sex, age group and geographic region as fixed factors and baseline measurement as a covariate. LS Mean Differences were calculated by subtracting Solifenacin 5 mg/Placebo from the comparison treatment group; Test type: Superiority or Other; p = 0.062, ANCOVA; LS Mean Difference = -0.68, 95% CI 2-sided [-1.40 to 0.03], Standard Error of Mean 0.366
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.91, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.63 to 0.56], Standard Error of Mean 0.302
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.20, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.98 to 0.20], Standard Error of Mean 0.302
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.96, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.62 to 0.58], Standard Error of Mean 0.305
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = -0.80, 95% CI 2-sided [-1.39 to -0.22], Standard Error of Mean 0.300
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.016, ANCOVA; LS Mean Difference = -0.88, 95% CI 2-sided [-1.59 to -0.16], Standard Error of Mean 0.363
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-1.68 to -0.27], Standard Error of Mean 0.360
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.91, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.87 to 0.77], Standard Error of Mean 0.417
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.76, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.94 to 0.69], Standard Error of Mean 0.415
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.99, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.82 to 0.81], Standard Error of Mean 0.416
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.77, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.82 to 0.60], Standard Error of Mean 0.361
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.058, ANCOVA; LS Mean Difference = -0.79, 95% CI 2-sided [-1.61 to 0.03], Standard Error of Mean 0.417
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.69, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.85 to 0.57], Standard Error of Mean 0.362
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.17, ANCOVA; LS Mean Difference = -0.50, 95% CI 2-sided [-1.21 to 0.21], Standard Error of Mean 0.362
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.73, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.84 to 0.59], Standard Error of Mean 0.364
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.012, ANCOVA; LS Mean Difference = -0.91, 95% CI 2-sided [-1.62 to -0.20], Standard Error of Mean 0.361
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.018, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-1.80 to -0.17], Standard Error of Mean 0.414
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.009, ANCOVA; LS Mean Difference = -1.08, 95% CI 2-sided [-1.89 to -0.28], Standard Error of Mean 0.412

3. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Incontinence Episodes Per 24 Hours
Description: The average number of incontinence episodes (any involuntary leakage of urine) per day was derived from the number of incontinence episodes recorded by the participant in the micturition diary for 3-days before the Baseline and Week 12 clinic visits.
Time Frame: Baseline and Week 12
Population: The Full Analysis Set-Incontinence comprised participants in the FAS who reported at least 1 incontinence episode in the baseline diary. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 17 | 13 | 18 | 15 | 35 | 15 | 35 | 33 | 32 | 24 | 24 | 20
incontinence episodes | -0.95 (0.365) | -0.74 (0.415) | -0.90 (0.353) | -1.26 (0.386) | -0.88 (0.252) | -0.97 (0.386) | -0.75 (0.251) | -0.85 (0.260) | -1.22 (0.266) | -1.14 (0.306) | -0.27 (0.304) | -0.97 (0.333)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; The ANCOVA model including the 2 main factors mirabegron dose and solifenacin dose and their interaction, sex, age group and geographic region as fixed factors and Baseline measurement as a covariate was used to calculate point estimates and 95% confidence intervals (CI) for change from Baseline within each treatment group and for differences between combination treatment groups and solifenacin 5 mg as well as for differences between active treatment groups and placebo; Test type: Superiority or Other; p = 0.51, Stratified Rank ANCOVA — Statistical comparisons were made using 2-sided tests at the 0.05 significance level. No adjustment for multiple testing was performed; P-values are from pairwise comparisons of the combination/active treatment groups vs. solifenacin 5 mg/placebo within a stratified rank ANCOVA model; LS Mean Difference = -0.09, 95% CI 2-sided [-1.00 to 0.82], Standard Error of Mean 0.460
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.21, Stratified Rank ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.57 to 0.83], Standard Error of Mean 0.355
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.89, Stratified Rank ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.68 to 0.74], Standard Error of Mean 0.361
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.001, Stratified Rank ANCOVA — P values were calculated from a pairwise comparison of the combination treatment groups vs solifenacin succinate 5 mg or placebo within the ANCOVA model; LS Mean Difference = -0.34, 95% CI 2-sided [-1.06 to 0.38], Standard Error of Mean 0.365
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.058, Stratified Rank ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-1.04 to 0.52], Standard Error of Mean 0.397
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.15, Stratified Rank ANCOVA; LS Mean Difference = 0.60, 95% CI 2-sided [-0.17 to 1.38], Standard Error of Mean 0.395
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.41, Stratified Rank ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.91 to 0.73], Standard Error of Mean 0.417
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.44, Stratified Rank ANCOVA; LS Mean Difference = 0.21, 95% CI 2-sided [-0.88 to 1.30], Standard Error of Mean 0.554
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.85, Stratified Rank ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.95 to 1.04], Standard Error of Mean 0.505
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.83, Stratified Rank ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-1.36 to 0.74], Standard Error of Mean 0.533
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.56, Stratified Rank ANCOVA; LS Mean Difference = 0.07, 95% CI 2-sided [-0.80 to 0.95], Standard Error of Mean 0.444
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.48, Stratified Rank ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-1.07 to 1.03], Standard Error of Mean 0.534
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.13, Stratified Rank ANCOVA; LS Mean Difference = 0.20, 95% CI 2-sided [-0.67 to 1.07], Standard Error of Mean 0.443
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.62, Stratified Rank ANCOVA; LS Mean Difference = 0.10, 2% CI 2-sided [-0.78 to 0.99], Standard Error of Mean 0.448
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.34, Stratified Rank ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-1.16 to 0.63], Standard Error of Mean 0.454
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.24, Stratified Rank ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-1.12 to 0.74], Standard Error of Mean 0.472
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.88, Stratified Rank ANCOVA; LS Mean Difference = 0.68, 95% CI 2-sided [-0.26 to 1.61], Standard Error of Mean 0.475
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.83, Stratified Rank ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.99 to 0.95], Standard Error of Mean 0.494

4. Secondary Outcome: Change From Baseline to Each Visit in Mean Volume Voided Per Micturition
Description: The average volume voided per micturition was calculated from the volume of each micturition measured by the participant and recorded in a micturition diary for 3 days before the Baseline and each post-baseline clinic visit.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full analysis set including participants with available data at Baseline and each post-baseline visit (indicated by "n")..
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
mL
  Week 2; n=80,71,76,74,148,73,145,145,136,141,76,77 | 8.7 (4.44) | 14.3 (4.71) | 26.0 (4.55) | 22.7 (4.62) | 23.1 (3.26) | 16.1 (4.64) | 22.5 (3.30) | 29.2 (3.30) | 29.9 (3.40) | 32.3 (3.34) | 29.5 (4.56) | 42.1 (4.52)
  Week 4; n=79,72,74,76,146,72,141,142,138,144,77,75 | 10.2 (4.93) | 16.8 (5.16) | 29.4 (5.09) | 24.8 (5.02) | 29.6 (3.63) | 28.3 (5.16) | 29.2 (3.69) | 36.5 (3.67) | 42.7 (3.73) | 44.5 (3.65) | 45.7 (5.00) | 54.5 (5.06)
  Week 8; n=77,70,73,75,147,73,143,142,134,143,76,74 | 13.5 (5.56) | 24.6 (5.83) | 35.4 (5.71) | 28.3 (5.63) | 30.1 (4.03) | 37.7 (5.71) | 35.6 (4.08) | 42.3 (4.09) | 49.7 (4.21) | 52.2 (4.08) | 55.8 (5.60) | 68.5 (5.67)
  Week 12;n=75,68,73,73,144,72,138,138,133,140,72,73 | 14.7 (6.12) | 23.0 (6.43) | 35.5 (6.20) | 36.9 (6.20) | 34.6 (4.42) | 35.8 (6.25) | 38.6 (4.52) | 43.7 (4.51) | 54.7 (4.60) | 56.6 (4.48) | 59.8 (6.26) | 66.2 (6.20)

5. Secondary Outcome: Change From Baseline to Each Visit in Mean Number of Micturitions Per 24 Hours
Description: The average number of micturitions (urinations) per 24 hours was derived from the number of urinations (excluding incontinence only episodes) per day recorded by the participant in the micturition diary for 3-days before the Baseline and each post-baseline clinic visit.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
micturitions
  Week 2; n=80,71,76,74,148,73,145,145,136,141,77,77 | -1.18 (0.240) | -1.69 (0.255) | -1.60 (0.246) | -1.49 (0.249) | -1.16 (0.176) | -1.32 (0.251) | -1.52 (0.178) | -1.95 (0.178) | -1.68 (0.184) | -2.21 (0.181) | -1.74 (0.244) | -2.35 (0.244)
  Week 4; n=79,72,74,76,147,73,141,142,138,144,77,75 | -1.68 (0.261) | -2.02 (0.273) | -1.99 (0.269) | -2.10 (0.266) | -1.80 (0.191) | -2.25 (0.271) | -2.03 (0.195) | -2.11 (0.194) | -2.29 (0.197) | -2.77 (0.193) | -2.55 (0.264) | -2.69 (0.267)
  Week 8; n=77,70,73,75,147,74,143,142,134,145,77,74 | -2.27 (0.270) | -2.27 (0.283) | -2.42 (0.277) | -2.46 (0.273) | -2.22 (0.196) | -2.97 (0.275) | -2.58 (0.198) | -2.66 (0.199) | -2.43 (0.205) | -3.20 (0.197) | -3.04 (0.270) | -3.49 (0.275)
  Week 12;n=75,69,73,73,144,73,138,138,133,144,75,73 | -2.59 (0.302) | -2.51 (0.314) | -2.67 (0.306) | -2.38 (0.306) | -2.58 (0.218) | -3.31 (0.306) | -2.64 (0.222) | -3.02 (0.222) | -2.64 (0.227) | -3.35 (0.218) | -3.47 (0.302) | -3.63 (0.306)

6. Secondary Outcome: Percentage of Participants With a Micturition Response
Description: A responder is defined as a participant with at most 8 micturitions per 24 hours post-baseline and a negative change (i.e. an improvement) from Baseline.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full analysis set participants with at least 8 micturitions per 24 hours at Baseline and including participants with available data at Baseline and each post-baseline visit (indicated by "n"); LOCF imputation was used for the End of Treatment (EOT) analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
percentage of participants
  Week 2; n=79,70,75,71,144,72,143,143,135,137,77,76 | 27.8 | 25.7 | 37.3 | 29.6 | 26.4 | 34.7 | 36.4 | 38.5 | 34.1 | 36.5 | 36.4 | 46.1
  Week 4; n=78,72,73,73,144,72,139,140,137,140,77,74 | 42.3 | 27.8 | 43.8 | 35.6 | 34.0 | 44.4 | 45.3 | 42.1 | 48.2 | 56.4 | 48.1 | 41.9
  Week 8; n=76,70,73,72,145,73,141,140,133,142,77,73 | 53.9 | 35.7 | 50.7 | 43.1 | 40.0 | 56.2 | 46.8 | 54.3 | 49.6 | 56.3 | 57.1 | 64.4
  Week 12;n=74,69,72,69,142,72,136,136,132,142,75,72 | 55.4 | 46.4 | 47.2 | 53.6 | 47.9 | 55.6 | 55.1 | 55.1 | 53.8 | 62.0 | 65.3 | 61.1
  EOT; n=79,75,76,73,146,75,144,145,140,146,78,79 | 53.2 | 42.7 | 47.4 | 54.8 | 47.9 | 54.7 | 54.2 | 53.1 | 52.1 | 61.6 | 65.4 | 58.2
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; All statistical comparisons are for End of Treatment using 2-sided tests at the 0.05 significance level. No adjustment for multiple testing was performed. The logistic regression model includes the 2 main factors mirabegron dose and solifenacin dose and their interaction, sex, age group and geographic region as fixed factors and baseline measurement as a covariate; Test type: Superiority or Other; p = 0.42, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.69 to 2.39]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.48, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.72 to 2.00]
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.69, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.67 to 1.83]
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.95, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.61 to 1.69]
Statistical Analysis 5: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.015, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [1.14 to 3.21]
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.11 to 3.84]
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.16, Regression, Logistic; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.84 to 2.84]
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.73, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.45 to 1.76]
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.70, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.45 to 1.72]
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.26, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.74 to 2.99]
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.69, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.63 to 2.04]
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.29, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.73 to 2.89]
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.31, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.75 to 2.45]
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.45, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.70 to 2.25]
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.64, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.64 to 2.07]
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.013, Regression, Logistic; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.18 to 3.94]
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.017, Regression, Logistic; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.16 to 4.66]
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.11, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.88 to 3.45]

7. Secondary Outcome: Change From Baseline to Each Visit in Mean Number of Incontinence Episodes Per 24 Hours
Description: The average number of incontinence episodes (any involuntary leakage of urine) per day was derived from the number of incontinence episodes recorded by the participant in the micturition diary for 3-days before the Baseline and each post-baseline clinic visit.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full Analysis Set-Incontinence including participants with available data at Baseline and each post-baseline visit (indicated by "n").
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 17 | 13 | 18 | 15 | 35 | 15 | 35 | 33 | 32 | 24 | 24 | 19
incontinence episodes
  Week 2; n=17,13,18,15,33,14,35,33,32,21,24,19 | -0.83 (0.168) | -0.43 (0.191) | -0.85 (0.162) | -0.98 (0.178) | -0.67 (0.119) | -0.71 (0.184) | -0.49 (0.116) | -0.64 (0.120) | -0.70 (0.122) | -0.65 (0.150) | -1.14 (0.140) | -0.77 (0.157)
  Week 4; n=17,10,18,15,34,14,34,30,32,23,24,19 | -0.87 (0.146) | -0.48 (0.189) | -0.89 (0.141) | -1.20 (0.155) | -0.80 (0.102) | -0.84 (0.160) | -0.73 (0.102) | -0.67 (0.109) | -0.81 (0.106) | -0.88 (0.125) | -1.18 (0.122) | -0.71 (0.137)
  Week 8; n=17,10,18,14,34,15,35,30,32,22,24,20 | -0.82 (0.163) | -0.65 (0.210) | -0.92 (0.157) | -1.12 (0.178) | -0.72 (0.114) | -1.04 (0.172) | -0.78 (0.112) | -0.82 (0.122) | -1.01 (0.118) | -0.95 (0.142) | -0.93 (0.136) | -0.91 (0.149)
  Week 12; n=17,10,18,13,34,14,33,30,30,23,24,20 | -0.93 (0.373) | -0.59 (0.482) | -0.89 (0.361) | -1.21 (0.424) | -0.84 (0.261) | -0.95 (0.409) | -0.74 (0.265) | -0.88 (0.279) | -1.20 (0.280) | -1.11 (0.319) | -0.27 (0.311) | -0.96 (0.341)

8. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes Post-baseline
Description: The percentage of participants with no incontinence episodes for the 3 days prior to each clinic visit derived from the micturition diary recorded by the participant.
Time Frame: Weeks 2, 4, 8 and 12
Population: Full Analysis Set-Incontinence including participants with available data at Baseline and each post-baseline visit (indicated by "n"); LOCF imputation was used for the End of Treatment (EOT) analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 17 | 13 | 18 | 15 | 35 | 15 | 35 | 33 | 32 | 24 | 24 | 20
percentage of participants
  Week 2; n=17,13,18,15,33,14,35,33,32,21,24,19 | 47.1 | 23.1 | 44.4 | 40.0 | 45.5 | 50.0 | 40.0 | 51.5 | 65.6 | 52.4 | 70.8 | 52.6
  Week 4; n=17,10,18,15,34,14,34,30,32,23,24,19 | 64.7 | 20.0 | 55.6 | 73.3 | 64.7 | 71.4 | 55.9 | 46.7 | 62.5 | 52.2 | 79.2 | 52.6
  Week 8; n=17,10,18,14,34,15,35,30,32,22,24,20 | 58.8 | 50.0 | 61.1 | 71.4 | 50.0 | 73.3 | 54.3 | 50.0 | 71.9 | 77.3 | 79.2 | 65.0
  Week 12; n=17,10,18,13,34,14,33,30,30,23,24,20 | 82.4 | 50.0 | 61.1 | 69.2 | 58.8 | 57.1 | 51.5 | 63.3 | 86.7 | 87.0 | 79.2 | 75.0
  EOT; n=17,13,18,15,35,15,35,33,32,24,24,20 | 82.4 | 46.2 | 61.1 | 66.7 | 60.0 | 53.3 | 54.3 | 60.6 | 87.5 | 87.5 | 79.2 | 75.0
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.52, Regression, Logistic; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.16 to 2.56]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.48, Regression, Logistic; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.23 to 1.99]
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.93, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.32 to 2.81]
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.013, Regression, Logistic; Odds Ratio (OR) = 6.12, 95% CI 2-sided [1.47 to 25.60]
Statistical Analysis 5: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.031, Regression, Logistic; Odds Ratio (OR) = 5.49, 95% CI 2-sided [1.17 to 25.77]
Statistical Analysis 6: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.059, Regression, Logistic; Odds Ratio (OR) = 3.84, 95% CI 2-sided [0.95 to 15.58]
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.36, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.48 to 7.58]
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.26, Regression, Logistic; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.05 to 2.17]
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.33, Regression, Logistic; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.08 to 2.31]
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.94, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.17 to 6.68]
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.29, Regression, Logistic; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.09 to 2.02]
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.15, Regression, Logistic; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.05 to 1.60]
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.11, Regression, Logistic; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.06 to 1.34]
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.26, Regression, Logistic; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.09 to 1.89]
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.28, Regression, Logistic; Odds Ratio (OR) = 2.67, 95% CI 2-sided [0.44 to 16.17]
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.36, Regression, Logistic; Odds Ratio (OR) = 2.39, 95% CI 2-sided [0.37 to 15.46]
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.56, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.29 to 9.72]
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.84, Regression, Logistic; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.15 to 4.76]

9. Secondary Outcome: Percentage of Participants With 50% Reduction in Incontinence Episodes
Description: The percentage of participants with at least a 50% decrease from Baseline in mean number of incontinence episodes per 24 hours during the 3 days prior to each clinic visit derived from the participant's micturition diary.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 17 | 13 | 18 | 15 | 35 | 15 | 35 | 33 | 32 | 24 | 24 | 20
percentage of participants
  Week 2; n=17,13,18,15,33,14,35,33,32,21,24,19 | 64.7 | 30.8 | 66.7 | 73.3 | 57.6 | 57.1 | 51.4 | 66.7 | 71.9 | 66.7 | 91.7 | 68.4
  Week 4; n=17,10,18,15,34,14,34,30,32,23,24,19 | 82.4 | 40.0 | 72.2 | 86.7 | 76.5 | 78.6 | 64.7 | 63.3 | 75.0 | 78.3 | 95.8 | 68.4
  Week 8; n=17,10,18,14,34,15,35,30,32,22,24,20 | 76.5 | 60.0 | 77.8 | 85.7 | 58.8 | 86.7 | 82.9 | 73.3 | 90.6 | 81.8 | 91.7 | 75.0
  Week 12; n=17,10,18,13,34,14,33,30,30,23,24,20 | 94.1 | 70.0 | 77.8 | 84.6 | 73.5 | 64.3 | 66.7 | 80.0 | 96.7 | 95.7 | 95.8 | 90.0
  EOT; n=17,13,18,15,35,15,35,33,32,24,24,20 | 94.1 | 61.5 | 77.8 | 86.7 | 74.3 | 66.7 | 68.6 | 75.8 | 96.9 | 95.8 | 95.8 | 90.0
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.48, Regression, Logistic; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.16 to 2.38]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.58, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.25 to 2.17]
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.93, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.34 to 3.28]
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 12.16, 95% CI 2-sided [1.40 to 105.30]
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.042, Regression, Logistic; Odds Ratio (OR) = 9.48, 95% CI 2-sided [1.08 to 83.24]
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.047, Regression, Logistic; Odds Ratio (OR) = 9.03, 95% CI 2-sided [1.03 to 79.19]
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.23, Regression, Logistic; Odds Ratio (OR) = 2.79, 95% CI 2-sided [0.52 to 14.90]
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.058, Regression, Logistic; Odds Ratio (OR) = 0.10, 95% CI 2-sided [0.01 to 1.08]
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.15, Regression, Logistic; Odds Ratio (OR) = 0.18, 95% CI 2-sided [0.02 to 1.87]
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.55, Regression, Logistic; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.04 to 5.99]
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.11, Regression, Logistic; Odds Ratio (OR) = 0.16, 95% CI 2-sided [0.02 to 1.48]
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.054, Regression, Logistic; Odds Ratio (OR) = 0.10, 95% CI 2-sided [0.01 to 1.05]
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.059, Regression, Logistic; Odds Ratio (OR) = 0.12, 95% CI 2-sided [0.01 to 1.08]
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.12, Regression, Logistic; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.02 to 1.58]
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.64, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.11 to 35.46]
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.76, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.09 to 27.42]
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.79, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.08 to 26.47]
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.55, Regression, Logistic; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.04 to 5.77]

10. Secondary Outcome: Change From Baseline to Each Visit in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: Urgency incontinence is the involuntary leakage of urine accompanied by or immediately preceded by urgency, and was derived from the number of incontinence episodes classified by the participant in a 3-day micturition diary as Grade 3 or 4 on the Patient Perception of Intensity of Urgency Scale: 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could postpone voiding a short while; 3 = Severe urgency, could not postpone voiding; 4 = Urge incontinence, leaked before arriving to the toilet.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full Analysis Set-Incontinence participants who had at least 1 urgency (grade 3 or 4) incontinence episode at Baseline, including participants with available data at Baseline and each post-baseline visit (indicated by "n"). LOCF was used for the End of Treatment (EOT) analysis.
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 17 | 13 | 18 | 15 | 35 | 15 | 35 | 33 | 32 | 24 | 24 | 20
urgency incontinence episodes
  Week 2; n=14,13,17,15,33,12,29,33,31,21,24,18 | -0.80 (0.178) | -0.59 (0.184) | -0.83 (0.161) | -0.96 (0.171) | -0.66 (0.115) | -0.77 (0.191) | -0.52 (0.123) | -0.68 (0.115) | -0.68 (0.120) | -0.64 (0.145) | -1.12 (0.135) | -0.76 (0.156)
  Week 4; n=14,10,17,15,34,12,28,30,31,22,24,18 | -0.83 (0.157) | -0.48 (0.185) | -0.93 (0.142) | -1.13 (0.151) | -0.77 (0.100) | -1.00 (0.169) | -0.73 (0.111) | -0.70 (0.107) | -0.81 (0.106) | -0.86 (0.125) | -1.20 (0.120) | -0.68 (0.138)
  Week 8; n=14,10,17,14,34,13,29,30,31,21,24,19 | -0.86 (0.173) | -0.65 (0.204) | -1.00 (0.157) | -1.04 (0.172) | -0.76 (0.110) | -1.16 (0.179) | -0.86 (0.119) | -0.84 (.118) | -0.99 (0.117) | -0.89 (0.141) | -0.91 (0.132) | -0.88 (0.148)
  Week 12; n=14,10,17,13,34,12,28,30,29,22,24,19 | -0.84 (0.420) | -0.54 (0.493) | -0.87 (0.379) | -1.13 (0.433) | -0.83 (0.267) | -1.13 (0.451) | -0.81 (0.295) | -0.91 (0.286) | -1.19 (0.292) | -1.06 (0.334) | -0.28 (0.319) | -0.93 (0.358)
  EOT; n=14,13,17,15,35,13,29,33,31,23,24,19 | -0.86 (0.411) | -0.80 (0.424) | -0.88 (0.372) | -1.17 (0.394) | -0.86 (0.258) | -1.13 (0.424) | -0.81 (0.283) | -0.87 (0.266) | -1.20 (0.277) | -1.08 (0.321) | -0.28 (0.312) | -0.94 (0.351)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; The ANCOVA model including the 2 main factors mirabegron dose and solifenacin dose and their interaction, sex, age group and geographic region as fixed factors and Baseline measurement as a covariate was used to calculate point estimates and 95% confidence intervals for change from Baseline within each treatment group and for differences between combination treatment groups and solifenacin 5 mg as well as for differences between active treatment groups and placebo; Test type: Superiority or Other; p = 0.25, Stratified Rank ANCOVA — All statistical comparisons are for change from Baseline to End of Treatment using 2-sided tests at the 0.05 significance level. No adjustment for multiple testing was performed; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -0.27, 95% CI 2-sided [-1.24 to 0.71], Standard Error of Mean 0.495
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.35, Stratified Rank ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.70 to 0.81], Standard Error of Mean 0.383
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 1.0, Stratified Rank ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.74 to 0.72], Standard Error of Mean 0.371
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.003, Stratified Rank ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-1.08 to 0.41], Standard Error of Mean 0.377
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.12, Stratified Rank ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-1.04 to 0.59], Standard Error of Mean 0.413
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.24, Stratified Rank ANCOVA; LS Mean Difference = 0.58, 95% CI 2-sided [-0.21 to 1.38], Standard Error of Mean 0.405
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.54, Stratified Rank ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.94 to 0.78], Standard Error of Mean 0.435
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.95, Stratified Rank ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-1.10 to 1.22], Standard Error of Mean 0.590
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.74, Stratified Rank ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-1.11 to 1.07], Standard Error of Mean 0.552
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.89, Stratified Rank ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-1.43 to 0.82], Standard Error of Mean 0.570
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.82, Stratified Rank ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.96 to 0.96], Standard Error of Mean 0.487
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.58, Stratified Rank ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-1.44 to 0.90], Standard Error of Mean 0.593
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.46, Stratified Rank ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.93 to 1.04], Standard Error of Mean 0.500
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.95, Stratified Rank ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.97 to 0.96], Standard Error of Mean 0.490
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.18, Stratified Rank ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-1.32 to 0.65], Standard Error of Mean 0.499
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.21, Stratified Rank ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-1.24 to 0.80], Standard Error of Mean 0.517
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.72, Stratified Rank ANCOVA; LS Mean Difference = 0.58, 95% CI 2-sided [-0.43 to 1.60], Standard Error of Mean 0.516
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.92, Stratified Rank ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-1.15 to 0.98], Standard Error of Mean 0.541

11. Secondary Outcome: Change From Baseline to Each Visit in Mean Number of Urgency Episodes (Grade 3 and/or 4) Per 24 Hours
Description: The average number of urgency episodes (the sudden, compelling desire to pass urine, which is difficult to defer), derived from urgency episodes classified by the participant in the 3-day micturition diary as grade 3 or 4 on the Patient Perception of Intensity of Urgency Scale: 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full analysis set including participants with available data at Baseline and each post-baseline visit (indicated by "n"). LOCF was used for the End of Treatment (EOT) analysis.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
urgency episodes
  Week 2; n=80,71,76,74,148,73,145,145,136,141,77,77 | -2.07 (0.276) | -2.06 (0.292) | -1.91 (0.282) | -2.49 (0.286) | -1.63 (0.202) | -1.97 (0.288) | -1.84 (0.205) | -2.59 (0.205) | -2.30 (0.211) | -2.57 (0.207) | -2.35 (0.281) | -2.23 (0.281)
  Week 4; n=79,72,74,76,147,73,141,142,138,144,77,75 | -2.55 (0.308) | -2.70 (0.322) | -2.70 (0.317) | -3.16 (0.313) | -2.24 (0.225) | -3.02 (0.320) | -2.64 (0.230) | -3.14 (0.229) | -3.08 (0.233) | -3.17 (0.228) | -3.04 (0.311) | -2.81 (0.316)
  Week 8; n=77,70,73,75,147,74,143,142,134,145,77,74 | -3.42 (0.318) | -2.86 (0.332) | -3.27 (0.325) | -3.61 (0.321) | -2.67 (0.229) | -3.63 (0.323) | -3.34 (0.232) | -3.60 (0.233) | -3.60 (0.240) | -3.85 (0.231) | -3.53 (0.317) | -3.63 (0.323)
  Week 12;n=75,69,73,73,144,73,138,138,133,144,75,73 | -3.69 (0.334) | -3.31 (0.347) | -3.65 (0.338) | -3.54 (0.338) | -2.71 (0.240) | -4.15 (0.337) | -3.26 (0.246) | -4.24 (0.246) | -3.98 (0.250) | -4.09 (0.240) | -3.76 (0.333) | -3.93 (0.338)
  EOT; n=80,76,77,77,150,76,146,147,141,150,78,80 | -3.53 (0.328) | -3.23 (0.336) | -3.44 (0.334) | -3.62 (0.334) | -2.73 (0.239) | -3.98 (0.336) | -3.21 (0.242) | -3.97 (0.242) | -3.86 (0.247) | -4.10 (0.239) | -3.71 (0.332) | -3.91 (0.327)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; All statistical comparisons are for change from Baseline to End of Treatment using 2-sided tests at the 0.05 significance level. No adjustment for multiple testing was performed. The ANCOVA model includes the 2 main factors mirabegron dose and solifenacin dose and their interaction, sex, age group and geographic region as fixed factors and baseline measurement as a covariate. LS Mean Differences were calculated by subtracting Solifenacin 5 mg/Placebo from the comparison treatment group; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -1.26, 95% CI 2-sided [-2.06 to -0.45], Standard Error of Mean 0.412
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.16, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-1.15 to 0.19], Standard Error of Mean 0.340
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.24, 95% CI 2-sided [-1.91 to -0.57], Standard Error of Mean 0.340
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -1.13, 95% CI 2-sided [-1.80 to -0.46], Standard Error of Mean 0.343
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.37, 95% CI 2-sided [-2.03 to -0.70], Standard Error of Mean 0.338
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.017, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-1.78 to -0.18], Standard Error of Mean 0.409
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -1.18, 95% CI 2-sided [-1.98 to -0.39], Standard Error of Mean 0.405
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.53, ANCOVA; LS Mean Difference = 0.29, 95% CI 2-sided [-0.63 to 1.22], Standard Error of Mean 0.469
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.85, ANCOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.83 to 1.01], Standard Error of Mean 0.468
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.84, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-1.01 to 0.83], Standard Error of Mean 0.468
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.050, ANCOVA; LS Mean Difference = 0.80, 95% CI 2-sided [-0.00 to 1.59], Standard Error of Mean 0.406
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.33, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-1.38 to 0.46], Standard Error of Mean 0.469
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.44, ANCOVA; LS Mean Difference = 0.32, 95% CI 2-sided [-0.48 to 1.12], Standard Error of Mean 0.407
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.28, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-1.24 to 0.36], Standard Error of Mean 0.408
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.42, ANCOVA; LS Mean Difference = -0.33, 95% CI 2-sided [-1.14 to 0.47], Standard Error of Mean 0.410
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.16, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-1.37 to 0.23], Standard Error of Mean 0.406
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.70, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-1.10 to 0.73], Standard Error of Mean 0.467
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.40, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-1.30 to 0.52], Standard Error of Mean 0.464

12. Secondary Outcome: Change From Baseline to Each Visit in Mean Level of Urgency
Description: Average of participants' ratings on the degree of urgency associated with each micturition and/or incontinence episode recorded in the 3-day micturition diary according to the Patient Perception of Intensity of Urgency Scale: 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
units on a scale
  Week 2; n=80,71,76,74,148,73,145,145,136,141,77,77 | -0.24 (0.043) | -0.19 (0.046) | -0.15 (0.044) | -0.25 (0.045) | -0.14 (0.032) | -0.21 (0.045) | -0.19 (0.032) | -0.26 (0.032) | -0.26 (0.033) | -0.28 (0.033) | -0.31 (0.044) | -0.20 (0.044)
  Week 4; n=79,72,74,76,147,73,141,142,138,144,77,75 | -0.32 (0.052) | -0.28 (0.054) | -0.26 (0.053) | -0.33 (0.053) | -0.23 (0.038) | -0.35 (0.054) | -0.32 (0.039) | -0.35 (0.039) | -0.35 (0.039) | -0.37 (0.038) | -0.41 (0.052) | -0.31 (0.053)
  Week 8; n=77,70,73,75,147,74,143,142,134,145,77,74 | -0.42 (0.059) | -0.30 (0.062) | -0.36 (0.061) | -0.45 (0.060) | -0.30 (0.043) | -0.44 (0.60) | -0.39 (0.043) | -0.41 (0.044) | -0.45 (0.045) | -0.46 (0.043) | -0.53 (0.059) | -0.43 (0.060)
  Week 12;n=75,69,73,73,144,73,138,138,133,144,75,73 | -0.48 (0.064) | -0.35 (0.067) | -0.44 (0.065) | -0.42 (0.065) | -0.33 (0.046) | -0.49 (0.065) | -0.43 (0.047) | -0.54 (0.047) | -0.50 (0.048) | -0.54 (0.046) | -0.61 (0.064) | -0.49 (0.065)
  EOT; n=80,76,77,77,150,76,146,147,141,150,78,80 | -0.46 (0.063) | -0.33 (0.064) | -0.41 (0.064) | -0.45 (0.064) | -0.33 (0.064) | -0.47 (0.064) | -0.42 (0.046) | -0.50 (0.046) | -0.48 (0.047) | -0.55 (0.046) | -0.59 (0.063) | -0.47 (0.063)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.062, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.30 to 0.01], Standard Error of Mean 0.079
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.15, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.22 to 0.03], Standard Error of Mean 0.065
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.30 to -0.05], Standard Error of Mean 0.065
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.017, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.29 to -0.03], Standard Error of Mean 0.066
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.35 to -0.10], Standard Error of Mean 0.065
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.41 to -0.11], Standard Error of Mean 0.078
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.070, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.29 to 0.01], Standard Error of Mean 0.077
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.15, ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.05 to 0.31], Standard Error of Mean 0.090
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.57, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.12 to 0.23], Standard Error of Mean 0.089
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.89, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.16 to 0.19], Standard Error of Mean 0.089
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.086, ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.02 to 0.29], Standard Error of Mean 0.077
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.88, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.19 to 0.16], Standard Error of Mean 0.090
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.61, ANCOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-0.11 to 0.19], Standard Error of Mean 0.078
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.58, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.20 to 0.11], Standard Error of Mean 0.078
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.76, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.18 to 0.13], Standard Error of Mean 0.078
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.23, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.25 to 0.06], Standard Deviation 0.077
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.15, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.30 to 0.05], Standard Error of Mean 0.089
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.94, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.18 to 0.17], Standard Error of Mean 0.088

13. Secondary Outcome: Change From Baseline to Each Visit in Mean Number of Pads Used Per 24 Hours
Description: The average number of times a participant recorded a new pad used per day during the 3-day micturition diary period.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full analysis set participants who had at least one use of pad at baseline, and including participants with available data at Baseline and each post-baseline visit (indicated by "n"). LOCF was used for the End of Treatment (EOT) analysis.
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
pads
  Week 2; n=33,33,34,31,74,23,62,55,62,62,45,30 | -0.81 (0.212) | -0.87 (0.212) | -0.88 (0.209) | -1.31 (0.219) | -0.92 (0.142) | -0.91 (0.255) | -0.86 (0.155) | -0.96 (0.164) | -0.89 (0.155) | -1.02 (0.155) | -1.13 (0.182) | -1.31 (0.223)
  Week 4; n=32,31,35,31,75,23,61,52,64,62,45,30 | -0.76 (0.224) | -0.93 (0.228) | -0.70 (0.214) | -1.62 (0.228) | -1.26 (0.147) | -1.23 (0.265) | -0.94 (0.162) | -1.09 (0.176) | -1.24 (0.159) | -1.30 (0.161) | -1.35 (0.189) | -1.36 (0.231)
  Week 8; n=30,31,34,31,74,24,63,52,64,61,45,30 | -0.97 (0.226) | -0.90 (0.223) | -1.11 (0.213) | -1.47 (0.223) | -1.25 (0.144) | -1.53 (0.253) | -1.10 (0.156) | -1.39 (0.172) | -1.29 (0.155) | -1.51 (0.159) | -1.37 (0.185) | -1.56 (0.227)
  Week 12; n=30,31,34,29,72,23,60,52,63,62,45,31 | -0.92 (0.246) | -0.97 (0.242) | -0.93 (0.231) | -1.35 (0.251) | -1.39 (0.159) | -1.75 (0.282) | -1.02 (0.174) | -1.44 (0.187) | -1.45 (0.170) | -1.63 (0.172) | -1.60 (0.201) | -1.60 (0.243)
  EOT; n=33,34,35,32,76,24,63,56,64,65,46,32 | -0.63 (0.244) | -1.04 (0.241) | -0.95 (0.237) | -1.44 (0.248) | -1.38 (0.161) | -1.73 (0.287) | -1.04 (0.177) | -1.38 (0.188) | -1.46 (0.176) | -1.63 (0.174) | -1.59 (0.207) | -1.63 (0.248)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.29, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.99 to 0.30], Standard Error of Mean 0.330
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.15, ANCOVA; LS Mean Difference = 0.35, 95% CI 2-sided [-0.12 to 0.82], Standard Error of Mean 0.239
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.99, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.48 to 0.49], Standard Error of Mean 0.248
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.76, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.54 to 0.40], Standard Error of Mean 0.239
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.30, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.71 to 0.22], Standard Error of Mean 0.238
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.43, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.72 to 0.31], Standard Error of Mean 0.262
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.40, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.83 to 0.33], Standard Error of Mean 0.296
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.24, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-1.08 to 0.27], Standard Error of Mean 0.343
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.36, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.98 to 0.36], Standard Error of Mean 0.340
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.020, ANCOVA; LS Mean Difference = -0.81, 95% CI 2-sided [-1.49 to -0.13], Standard Error of Mean 0.348
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.011, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.33 to -0.18], Standard Error of Mean 0.293
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -1.10, 95% CI 2-sided [-1.84 to -0.36], Standard Error of Mean 0.377
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.18, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-1.00 to 0.19], Standard Error of Mean 0.301
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.015, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.35 to -0.14], Standard Error of Mean 0.308
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.006, ANCOVA; LS Mean Difference = -0.82, 95% CI 2-sided [-1.41 to -0.23], Standard Error of Mean 0.301
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.00, 95% CI 2-sided [-1.59 to -0.41], Standard Error of Mean 0.300
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.96, 95% CI 2-sided [-1.59 to -0.33], Standard Error of Mean 0.320
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -1.00, 95% CI 2-sided [-1.68 to -0.31], Standard Error of Mean 0.348

14. Secondary Outcome: Change From Baseline to Each Visit in Mean Number of Nocturia Episodes Per 24-Hours
Description: Nocturia is defined as waking at night one or more times to void. The average number of times a participant urinated (excluding incontinence only episodes) during sleeping time per day was derived from the 3-day micturition diary.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full analysis set participants who had at least one nocturia episode at baseline, and including participants with available data at Baseline and each post-baseline visit (indicated by "n"). LOCF was used for the End of Treatment (EOT) analysis.
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
nocturia episodes
  Week 2; n=78,69,75,72,144,71,142,138,133,138,74,73 | -0.33 (0.115) | -0.37 (0.123) | -0.60 (0.118) | -0.38 (0.120) | -0.30 (0.085) | -0.45 (0.121) | -0.43 (0.086) | -0.51 (0.087) | -0.49 (0.088) | -0.61 (0.087) | -0.43 (0.119) | -0.53 (0.119)
  Week 4; n=77,69,74,74,143,71,138,135,134,141,74,71 | -0.50 (0.116) | -0.60 (0.123) | -0.71 (0.118) | -0.55 (0.118) | -0.47 (0.085) | -0.74 (0.121) | -0.59 (0.087) | -0.54 (0.088) | -0.69 (0.088) | -0.80 (0.086) | -0.67 (0.119) | -0.75 (0.121)
  Week 8; n=75,67,73,73,143,72,140,135,130,142,74,70 | -0.64 (0.126) | -0.65 (0.133) | -0.68 (0.127) | -0.80 (0.127) | -0.65 (0.091) | -1.01 (0.128) | -0.76 (0.092) | -0.79 (0.094) | -0.76 (0.095) | -0.98 (0.091) | -0.81 (0.127) | -0.91 (0.130)
  Week 12;n=73,66,73,71,140,71,135,131,130,141,72,69 | -0.79 (0.146) | -0.69 (0.154) | -0.84 (0.146) | -0.59 (0.148) | -0.70 (0.106) | -0.99 (0.148) | -0.75 (0.108) | -0.81 (0.109) | -0.80 (0.110) | -1.05 (0.105) | -0.98 (0.147) | -1.03 (0.150)
  EOT; n=78,73,76,75,146,74,143,140,137,147,75,76 | -0.74 (0.140) | -0.69 (0.145) | -0.82 (0.142) | -0.68 (0.143) | -0.69 (0.102) | -0.95 (0.144) | -0.73 (0.104) | -0.77 (0.105) | -0.77 (0.106) | -1.04 (0.102) | -0.94 (0.143) | -0.96 (0.142)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.15, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.60 to 0.09], Standard Error of Mean 0.177
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.78, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.33 to 0.25], Standard Error of Mean 0.146
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.58, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.37 to 0.21], Standard Error of Mean 0.146
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.60, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.37 to 0.21], Standard Error of Mean 0.147
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.017, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.63 to -0.06], Standard Error of Mean 0.145
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.16, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.60 to 0.10], Standard Error of Mean 0.176
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.13, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.61 to 0.08], Standard Error of Mean 0.175
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.81, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.35 to 0.44], Standard Error of Mean 0.201
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.67, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.48 to 0.31], Standard Error of Mean 0.199
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.77, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.33 to 0.45], Standard Error of Mean 0.200
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.81, ANCOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-0.30 to 0.38], Standard Error of Mean 0.81
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.30, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.60 to 0.18], Standard Error of Mean 0.201
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.99, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.34 to 0.34], Standard Error of Mean 0.174
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.82, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.38 to 0.30], Standard Error of Mean 0.175
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.84, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.38 to 0.31], Standard Error of Mean 0.175
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.080, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.64 to 0.04], Standard Error of Mean 0.173
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.30, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.60 to 0.18], Standard Error of Mean 0.200
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.26, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.62 to 0.17], Standard Error of Mean 0.199

15. Secondary Outcome: Change From Baseline to End of Treatment in Patient Perception of Bladder Condition (PPBC)
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. A negative change from Baseline score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full Analysis Set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 78 | 73 | 76 | 75 | 147 | 73 | 141 | 143 | 136 | 144 | 76 | 78
units on a scale | -1.4 (0.14) | -1.4 (0.14) | -1.5 (0.14) | -1.5 (0.14) | -1.3 (0.10) | -1.5 (0.14) | -1.4 (0.10) | -1.7 (0.10) | -1.7 (0.10) | -1.8 (0.10) | -1.8 (0.14) | -1.6 (0.14)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.38, ANCOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.85, ANCOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.3 to 0.3], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.024, ANCOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to -0.0], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.14
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.17
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.15, ANCOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.17
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.99, ANCOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.4], Standard Error of Mean 0.20
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.67, ANCOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.19
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.44, ANCOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.19
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.88, ANCOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.53, ANCOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.20
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 1.0, ANCOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.3 to 0.3], Standard Error of Mean 0.17
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.084, ANCOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.17
Statistical Analysis 15: Comparison: Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.030, ANCOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.0], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.020, ANCOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.17
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.017, ANCOVA; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.1], Standard Error of Mean 0.19
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.26, ANCOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.2], Standard Error of Mean 0.19

16. Secondary Outcome: Percentage of Participants With Improvement in PPBC
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. Improvement was defined as at least a 1-point improvement (decrease) from Baseline in PPBC score.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 78 | 73 | 76 | 75 | 147 | 73 | 141 | 143 | 136 | 144 | 76 | 78
percentage of participants | 69.2 | 76.7 | 78.9 | 68.0 | 72.8 | 84.9 | 74.5 | 83.2 | 77.9 | 82.6 | 82.9 | 75.6
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.040, Regression, Logistic; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.04 to 4.95]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.73, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.63 to 1.92]
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.050, Regression, Logistic; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.00 to 3.30]
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.21, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.81 to 2.59]
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.021, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.11 to 3.66]
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.19, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.79 to 3.40]
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.74, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.57 to 2.19]
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.57, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.58 to 2.71]
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.19, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.77 to 3.64]
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.69, Regression, Logistic; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.41 to 1.79]
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.90, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.55 to 1.99]
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.048, Regression, Logistic; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.01 to 5.55]
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.67, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.60 to 2.22]
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.070, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.95 to 3.78]
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.23, Regression, Logistic; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.77 to 2.98]
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.034, Regression, Logistic; Odds Ratio (OR) = 2.11, 95% CI 2-sided [1.06 to 4.19]
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.20, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.76 to 3.84]
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.68, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.55 to 2.49]

17. Secondary Outcome: Percentage of Participants With Major Improvement in PPBC
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. Major improvement was defined as at least a 2-point improvement (decrease) from Baseline in PPBC score.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 78 | 73 | 76 | 75 | 147 | 73 | 141 | 143 | 136 | 144 | 76 | 78
percentage of participants | 39.7 | 42.5 | 38.2 | 44.0 | 42.2 | 46.6 | 48.2 | 52.4 | 54.4 | 54.9 | 57.9 | 50.0
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.62, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.64 to 2.12]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.25, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.82 to 2.17]
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.11, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.91 to 2.41]
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.020, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.10 to 2.97]
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.15 to 3.05]
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.072, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.95 to 3.10]
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.29, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.77 to 2.44]
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.94, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.49 to 1.93]
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.80, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.46 to 1.81]
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.67, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.59 to 2.28]
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.55 to 1.80]
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.66, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.59 to 2.31]
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.35, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.73 to 2.40]
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.19, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.82 to 2.67]
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.054, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.99 to 3.28]
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.038, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.04 to 3.38]
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.12, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.87 to 3.39]
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.36, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.70 to 2.67]

18. Secondary Outcome: Percentage of Participants With Deterioration in PPBC
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. Deterioration was defined as at least a 1 point increase from Baseline in PPBC score.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 78 | 73 | 76 | 75 | 147 | 73 | 141 | 143 | 136 | 144 | 76 | 78
percentage of participants | 6.4 | 4.1 | 5.3 | 4.0 | 4.8 | 2.7 | 4.3 | 2.8 | 2.9 | 1.4 | 1.3 | 6.4
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.32, Regression, Logistic; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.06 to 2.43]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.65, Regression, Logistic; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.21 to 2.61]
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.39, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.13 to 2.19]
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.22, Regression, Logistic; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.10 to 1.67]
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.082, Regression, Logistic; Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.04 to 1.22]
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.36, Regression, Logistic; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.04 to 3.20]
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.51, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.42 to 5.71]
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.99, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.19 to 5.36]
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.96, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.24 to 4.59]
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.57, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.12 to 3.30]
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.93, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.28 to 3.95]
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.37, Regression, Logistic; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.06 to 2.79]
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.74, Regression, Logistic; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.20 to 3.13]
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.46, Regression, Logistic; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.12 to 2.59]
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.28, Regression, Logistic; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.10 to 1.96]
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.11, Regression, Logistic; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.04 to 1.40]
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.40, Regression, Logistic; Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.04 to 3.66]
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.50, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.39 to 6.85]

19. Secondary Outcome: Change From Baseline to End of Treatment in Symptom Bother Score as Assessed by the Overactive Bladder Questionnaire (OAB-q)
Description: Overactive bladder symptoms were assessed using the symptom bother scale of the overactive bladder questionnaire. The symptom bother scale consists of 8 questions answered by the participant on a scale from 1-6. The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 to 100, with 100 indicating worst severity. A negative change from Baseline in symptom bother score indicates improvements.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 79 | 75 | 76 | 77 | 150 | 75 | 144 | 145 | 139 | 146 | 78 | 78
units on a scale | -25.5 (1.96) | -27.1 (2.01) | -27.5 (2.00) | -29.8 (1.99) | -26.8 (1.42) | -29.9 (2.01) | -28.0 (1.45) | -31.7 (1.45) | -32.0 (1.48) | -33.5 (1.44) | -33.6 (1.97) | -31.4 (1.97)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.21, ANCOVA; LS Mean Difference = -3.1, 95% CI 2-sided [-8.0 to 1.7], Standard Error of Mean 2.47
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.54, ANCOVA; LS Mean Difference = -1.3, 95% CI 2-sided [-5.2 to 2.7], Standard Error of Mean 2.03
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.016, ANCOVA; LS Mean Difference = -4.9, 95% CI 2-sided [-8.9 to -0.9], Standard Error of Mean 2.03
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.011, ANCOVA; LS Mean Difference = -5.2, 95% CI 2-sided [-9.3 to -1.2], Standard Error of Mean 2.05
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -6.7, 95% CI 2-sided [-10.7 to -2.8], Standard Error of Mean 2.03
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = -6.8, 95% CI 2-sided [-11.6 to -2.0], Standard Error of Mean 2.43
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.056, ANCOVA; LS Mean Difference = -4.7, 95% CI 2-sided [-9.4 to 0.1], Standard Error of Mean 2.44
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.56, ANCOVA; LS Mean Difference = -1.6, 95% CI 2-sided [-7.1 to 3.9], Standard Error of Mean 2.81
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.48, ANCOVA; LS Mean Difference = -2.0, 95% CI 2-sided [-7.5 to 3.5], Standard Error of Mean 2.80
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.13, ANCOVA; LS Mean Difference = -4.3, 95% CI 2-sided [-9.8 to 1.2], Standard Error of Mean 0.13
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.61, ANCOVA; LS Mean Difference = -1.2, 95% CI 2-sided [-6.0 to 3.5], Standard Error of Mean 2.42
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.12, ANCOVA; LS Mean Difference = -4.4, 95% CI 2-sided [-9.9 to 1.2], Standard Error of Mean 2.81
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.31, ANCOVA; LS Mean Difference = -2.5, 95% CI 2-sided [-7.3 to 2.3], Standard Error of Mean 2.44
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.012, ANCOVA; LS Mean Difference = -6.1, 95% CI 2-sided [-10.9 to -1.3], Standard Error of Mean 2.44
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = -6.5, 95% CI 2-sided [-11.3 to -1.7], Standard Error of Mean 2.46
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -8.0, 95% CI 2-sided [-12.8 to -3.2], Standard Error of Mean 2.44
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -8.0, 95% CI 2-sided [-13.5 to -2.6], Standard Error of Mean 2.78
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.035, ANCOVA; LS Mean Difference = -5.9, 95% CI 2-sided [-11.4 to -0.4], Standard Error of Mean 2.79

20. Secondary Outcome: Percentage of Participants With a Symptom Bother Response
Description: Overactive bladder symptoms were assessed using the symptom bother scale of the overactive bladder questionnaire. The symptom bother scale consists of 8 questions answered by the participant on a scale from 1-6. The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 to 100, with 100 indicating worst severity. Symptom bother response is defined as improvement (decrease) of at least 10 points from Baseline.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 79 | 75 | 76 | 77 | 150 | 75 | 144 | 145 | 139 | 146 | 78 | 78
percentage of participants | 73.4 | 84.0 | 78.9 | 85.7 | 81.3 | 85.3 | 82.6 | 85.5 | 85.6 | 88.4 | 88.5 | 83.3
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.40, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.63 to 3.20]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.89, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.55 to 1.97]
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.57, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.63 to 2.33]
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.36, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.70 to 2.66]
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.15, Regression, Logistic; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.83 to 3.32]
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.31, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.67 to 3.59]
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.81, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.42 to 1.95]
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.19, Regression, Logistic; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.75 to 4.08]
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.59, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.56 to 2.77]
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.13, Regression, Logistic; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.83 to 4.71]
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.20, Regression, Logistic; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.78 to 3.16]
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.070, Regression, Logistic; Odds Ratio (OR) = 2.24, 95% CI 2-sided [0.94 to 5.34]
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.17, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.81 to 3.33]
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.084, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.92 to 3.92]
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.043, Regression, Logistic; Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.02 to 4.48]
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.013, Regression, Logistic; Odds Ratio (OR) = 2.61, 95% CI 2-sided [1.22 to 5.58]
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.053, Regression, Logistic; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.99 to 5.97]
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.39, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.63 to 3.26]

21. Secondary Outcome: Change From Baseline to End of Treatment in Health-related Quality of Life (HRQL) Total Score
Description: Health-related quality of life was assessed by the HRQL subscales (coping, concern, sleep and social interaction) of the overactive bladder questionnaire (OABq). The HRQL total score was calculated by adding the 4 HRQL subscale scores, and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from Baseline in HRQL score indicates improvements.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 79 | 75 | 76 | 77 | 150 | 75 | 144 | 145 | 139 | 146 | 78 | 78
units on a scale | 24.5 (2.03) | 22.5 (2.08) | 25.8 (2.07) | 27.7 (2.05) | 23.7 (1.47) | 26.6 (2.08) | 25.5 (1.50) | 28.5 (1.50) | 29.2 (1.53) | 30.1 (1.49) | 30.3 (2.04) | 28.9 (2.04)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.26, ANCOVA; LS Mean Difference = 2.9, 95% CI 2-sided [-2.1 to 7.9], Standard Error of Mean 2.55
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.38, ANCOVA; LS Mean Difference = 1.8, 95% CI 2-sided [-2.3 to 6.0], Standard Error of Mean 2.10
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.022, ANCOVA; LS Mean Differrence = 4.8, 95% CI 2-sided [0.7 to 8.9], Standard Error of Mean 2.10
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.010, ANCOVA; LS Mean Difference = 5.5, 95% CI 2-sided [1.3 to 9.7], Standard Error of Mean 2.12
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = 6.4, 95% CI 2-sided [2.3 to 10.5], Standard Error of Mean 2.09
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = 6.7, 95% CI 2-sided [1.7 to 11.6], Standard Error of Mean 2.52
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.037, ANCOVA; LS Mean Difference = 5.3, 95% CI 2-sided [0.3 to 10.2], Standard Error of Mean 2.52
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.50, ANCOVA; LS Mean Difference = -2.0, 95% CI 2-sided [-7.7 to 3.7], Standard Error of Mean 2.90
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.65, ANCOVA; LS Mean Difference = 1.3, 95% CI 2-sided [-4.4 to 7.0], Standard Error of Mean 2.89
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.25, ANCOVA; LS Mean Difference = 3.3, 95% CI 2-sided [-2.4 to 8.9], Standard Error of Mean 2.88
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.76, ANCOVA; LS Mean Difference = -0.8, 95% CI 2-sided [-5.7 to 4.1], Standard Error of Mean 2.51
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.47, ANCOVA; LS Mean Difference = 2.1, 95% CI 2-sided [-3.6 to 7.8], Standard Error of Mean 2.91
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.67, ANCOVA; LS Mean Difference = 1.1, 95% CI 2-sided [-3.9 to 6.0], Standard Error of Mean 2.52
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.11, ANCOVA; LS Mean Difference = 4.0, 95% CI 2-sided [-0.9 to 9.0], Standard Error of Mean 2.52
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.062, ANCOVA; LS Mean Difference = 4.7, 95% CI 2-sided [-0.2 to 9.7], Standard Error of Mean 2.54
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.025, ANCOVA; LS Mean Difference = 5.6, 95% CI 2-sided [0.7 to 10.6], Standard Error of Mean 2.52
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.041, ANCOVA; LS Mean Difference = 5.9, 95% CI 2-sided [0.2 to 11.5], Standard Error of Mean 2.88
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.12, ANCOVA; LS Mean Difference = 4.5, 95% CI 2-sided [-1.2 to 10.1], Standard Error of Mean 2.88

22. Secondary Outcome: Percentage of Participants With a Health-related Quality of Life Total Score Response
Description: Health-related quality of life was assessed by the HRQL subscales (coping, concern, sleep and social interaction) of the overactive bladder questionnaire (OABq). The HRQL total score was calculated by adding the 4 HRQL subscale scores, and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. HRQL response is defined as improvement (decrease) of at least 10 points from Baseline.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 79 | 75 | 76 | 77 | 150 | 75 | 144 | 145 | 139 | 146 | 78 | 78
percentage of participants | 67.1 | 57.3 | 71.1 | 74.0 | 72.7 | 74.7 | 72.9 | 78.6 | 77.0 | 84.2 | 79.5 | 82.1
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; All statistical comparisons were made using 2-sided tests at the 0.05 significance level. No adjustment for multiple testing was performed. The logistic regression model includes the 2 main factors mirabegron dose and solifenacin dose and their interaction, sex, age group and geographic region as fixed factors and baseline measurement as a covariate; Test type: Superiority or Other; p = 0.92, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.52 to 2.08]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.98, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.58 to 1.77]
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.45, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.70 to 2.23]
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.24, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.79 to 2.53]
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.19 to 4.09]
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.32, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.70 to 2.90]
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.27, Regression, Logistic; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.72 to 3.14]
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.064, Regression, Logistic; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.24 to 1.04]
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.57, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.59 to 2.61]
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.55, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.59 to 2.68]
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.75, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.58 to 2.13]
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.72, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.53 to 2.49]
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.74, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.58 to 2.15]
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.34, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.71 to 2.71]
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.19, Regression, Logistic; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.80 to 3.07]
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 2.45, 95% CI 2-sided [1.22 to 4.94]
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.25, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.72 to 3.47]
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.21, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.74 to 3.75]

23. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) Mobility Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state:
  I have no problems in walking about; I have some problems in walking about; I am confined to bed.
  In the table below, each row title lists Baseline health status first followed by End of Treatment health status and reports the number of patients in that category.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
participants
  No problem → No problem | 60 | 58 | 63 | 59 | 118 | 54 | 94 | 113 | 102 | 120 | 59 | 56
  No problem → Some problems | 6 | 1 | 4 | 4 | 6 | 4 | 9 | 5 | 9 | 1 | 0 | 5
  No problem → Confined to bed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No problem → Missing data | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 2
  Some problems → No problems | 5 | 6 | 6 | 4 | 11 | 8 | 21 | 15 | 13 | 14 | 11 | 8
  Some problems → Some problems | 8 | 10 | 3 | 10 | 15 | 9 | 20 | 12 | 15 | 11 | 8 | 9
  Some problems → Confined to bed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Some problems → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Confined → No problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Confined → Some problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Confined → Confined to bed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Confined → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → No problem | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
  Missing data → Some problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Missing data → Confined to bed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) Self-care Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state:
  I have no problems with self-care; I have some problems washing or dressing myself; I am unable to wash or dress myself.
  In the table below, each row title lists Baseline health status first followed by End of Treatment health status and reports the number of patients in that category.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
participants
  No problem → No problem | 76 | 69 | 73 | 72 | 138 | 68 | 128 | 138 | 130 | 141 | 74 | 72
  No problem → Some problems | 0 | 1 | 3 | 2 | 2 | 2 | 5 | 2 | 1 | 1 | 1 | 0
  No problem → Unable | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  No problem → Missing data | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 2
  Some problems → No problems | 1 | 4 | 0 | 1 | 6 | 3 | 8 | 3 | 3 | 2 | 1 | 2
  Some problems → Some problems | 2 | 1 | 0 | 2 | 3 | 1 | 3 | 2 | 4 | 2 | 2 | 4
  Some problems → Unable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Some problems → Missing data | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unable → No problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unable → Some problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unable → Unable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unable → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → No problem | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
  Missing data → Some problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Missing data → Unable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) Usual Activities Score
Description: The EQ-5D is a standardized, nondisease-specific instrument for describing health status. Participants were asked which statement best describes their health state with regard to usual activities (work, study or leisure): I have no problems performing my usual activities; I have some problems performing my usual activities; I am unable to perform my usual activities.
  In the table below, each row title lists Baseline health status first followed by End of Treatment health status and reports the number of patients in that category.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
participants
  No problem → No problem | 62 | 52 | 58 | 60 | 115 | 57 | 89 | 110 | 106 | 109 | 57 | 48
  No problem → Some problems | 2 | 2 | 3 | 2 | 3 | 4 | 8 | 3 | 9 | 4 | 1 | 5
  No problem → Unable | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  No problem → Missing data | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 2
  Some problems → No problems | 11 | 11 | 8 | 11 | 16 | 7 | 29 | 24 | 12 | 21 | 14 | 14
  Some problems → Some problems | 4 | 10 | 6 | 4 | 13 | 6 | 18 | 8 | 11 | 12 | 4 | 8
  Some problems → Unable | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Some problems → Missing data | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Unable → No problems | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Unable → Some problems | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Unable → Unable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unable → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → No problem | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
  Missing data → Some problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Missing data → Unable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) Pain/Discomfort Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state:
  I have no pain or discomfort; I have moderate pain or discomfort; I have extreme pain or discomfort. In the table below, each row title lists Baseline health status first followed by End of Treatment health status and reports the number of participants in that category.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
participants
  No pain → No pain | 38 | 33 | 40 | 38 | 70 | 35 | 67 | 61 | 66 | 73 | 39 | 32
  No pain → Moderate pain | 9 | 12 | 6 | 4 | 15 | 3 | 6 | 11 | 14 | 7 | 8 | 6
  No pain → Extreme pain | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  No pain → Missing data | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2
  Moderate pain → No pain | 12 | 14 | 10 | 12 | 24 | 13 | 24 | 34 | 28 | 36 | 14 | 20
  Moderate pain → Moderate pain | 16 | 15 | 19 | 19 | 37 | 18 | 37 | 33 | 27 | 25 | 12 | 18
  Moderate pain → Extreme pain | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 1 | 2
  Moderate pain → Missing data | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Extreme pain → No pain | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 1 | 1 | 1 | 0 | 0
  Extreme pain → Moderate pain | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 4 | 3 | 0
  Extreme pain → Extreme pain | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 2 | 1 | 0 | 1 | 0
  Extreme pain → Missing data | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → No pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Missing data → Moderate pain | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Missing data → Extreme pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) Anxiety/Depression Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state:
  I am not anxious or depressed; I am moderately anxious or depressed; I am extremely anxious or depressed. In the table below, each row title lists Baseline health status first followed by End of Treatment health status and reports the number of patients in that category.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
participants
  No anxiety → No anxiety | 41 | 38 | 39 | 42 | 76 | 36 | 81 | 78 | 76 | 80 | 44 | 36
  No anxiety → Moderate anxiety | 5 | 8 | 7 | 4 | 11 | 6 | 7 | 5 | 9 | 3 | 5 | 6
  No anxiety → Extreme anxiety | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  No anxiety → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2
  Moderate anxiety → No anxiety | 17 | 9 | 15 | 21 | 24 | 19 | 25 | 35 | 28 | 33 | 15 | 14
  Moderate anxiety → Moderate anxiety | 13 | 18 | 14 | 9 | 33 | 12 | 21 | 22 | 19 | 26 | 8 | 19
  Moderate anxiety → Extreme anxiety | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 1
  Moderate anxiety → Missing data | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
  Extreme anxiety → No anxiety | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 2 | 2 | 3 | 2
  Extreme anxiety → Moderate anxiety | 2 | 1 | 0 | 0 | 0 | 1 | 7 | 1 | 4 | 1 | 1 | 0
  Extreme anxiety → Extreme anxiety | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0
  Extreme anxiety → Missing data | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → No anxiety | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
  Missing data → Moderate anxiety | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data → Extreme anxiety | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Missing data → Missing data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Change From Baseline to End of Treatment in European Quality of Life-5 Dimensions (EQ-5D) Visual Analog Scale (VAS)
Description: The EQ-5D is an international, standardized, generic instrument for describing and evaluating health status. Health status is assessed by patients evaluating their health on a vertical, visual analog scale from 0 to 100 where the endpoints are labeled 'Worst imaginable health state' (=0) and 'Best imaginable health state' (=100). On the EQ-5D VAS, a positive change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 79 | 75 | 76 | 77 | 150 | 75 | 144 | 145 | 139 | 146 | 78 | 78
units on a scale | 13.1 (21.11) | 5.8 (19.38) | 14.3 (22.38) | 11.1 (19.26) | 11.9 (21.33) | 13.3 (21.81) | 11.6 (21.94) | 12.5 (19.95) | 11.8 (18.91) | 15.9 (20.94) | 15.3 (24.17) | 11.1 (23.18)

29. Secondary Outcome: Change From Baseline to End of Treatment in Work Productivity and Activity Impairment (WPAI)
Description: This 6-item assessment measures productivity losses during the past 7 days and includes measures on work time missed due to health, impairment while working due to health (the participant's assessment of the degree to which health affected their productivity while working), overall work impairment due to health (takes into account both hours missed due to health and the participant's assessment of the degree to which health affected their productivity while working) and activity impairment due to health (the degree in which health problems affected their ability to do regular daily activities). Scores for each measure are expressed from 0 to 100 with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 80 | 76 | 77 | 77 | 150 | 76 | 146 | 147 | 141 | 150 | 78 | 80
units on a scale
  Percent work time missed | -2.44 (10.580) | 0.53 (3.031) | -0.24 (1.988) | -2.85 (11.205) | -1.29 (12.606) | -0.28 (2.737) | -0.55 (12.816) | -0.83 (17.199) | -0.84 (5.330) | -1.65 (4.654) | 0.79 (6.757) | -1.12 (11.025)
  Percent impairment while working | -7.50 (24.539) | -16.13 (24.314) | -10.00 (22.220) | -16.67 (25.207) | -17.33 (22.689) | -10.00 (17.728) | -8.43 (27.523) | -17.72 (26.187) | -13.85 (27.664) | -13.39 (24.515) | -18.00 (29.642) | -9.29 (26.377)
  Percent overall work impairment | -9.50 (24.090) | -16.32 (24.653) | -9.91 (21.464) | -17.88 (28.134) | -17.26 (25.196) | -9.95 (17.988) | -8.59 (29.521) | -17.16 (27.695) | -14.00 (27.384) | -14.18 (25.092) | -17.69 (29.323) | -10.32 (27.580)
  Percent activity impairment | -9.62 (26.989) | -14.52 (27.439) | -13.95 (26.386) | -13.73 (27.052) | -14.38 (24.182) | -17.12 (27.813) | -14.11 (31.398) | -25.31 (26.158) | -17.43 (29.008) | -20.42 (27.094) | -19.34 (27.439) | -19.74 (30.021)

30. Secondary Outcome: Change From Baseline to End of Treatment in Treatment Satisfaction on Visual Analog Scale (TS-VAS)
Description: The TS-VAS is a visual analog scale (VAS) that asks patients to rate their satisfaction with treatment by placing a vertical mark on a 10 cm line where the endpoints are labeled 'No, not at all' on the left (=0) to 'Yes, completely satisfied' on the right (=10). A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available Baseline and post-baseline data; LOCF imputation was used
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Solifenacin 10 mg + Mirabegron 25 mg | Solifenacin 10 mg + Mirabegron 50 mg
Number analyzed (Participants) | 78 | 73 | 76 | 75 | 147 | 73 | 141 | 143 | 136 | 144 | 76 | 78
units on a scale | 2.44 (0.298) | 2.61 (0.307) | 3.17 (0.301) | 3.10 (0.303) | 2.78 (0.217) | 2.96 (0.307) | 2.96 (0.221) | 3.24 (0.220) | 3.47 (0.225) | 3.24 (0.219) | 3.51 (0.301) | 3.72 (0.297)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.63, ANCOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.56 to 0.92], Standard Error of Mean 0.376
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.56, ANCOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.43 to 0.79], Standard Error of Mean 0.310
Statistical Analysis 3: Comparison: Solifenacin 5 mg vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.14, ANCOVA; LS Mean Difference = 0.46, 95% CI 2-sided [-0.15 to 1.06], Standard Error of Mean 0.308
Statistical Analysis 4: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.027, ANCOVA; LS Mean Difference = 0.69, 95% CI 2-sided [0.08 to 1.30], Standard Error of Mean 0.313
Statistical Analysis 5: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.13, ANCOVA; LS Mean Difference = 0.46, 95% CI 2-sided [-0.14 to 1.07], Standard Error of Mean 0.308
Statistical Analysis 6: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.049, ANCOVA; LS Mean Difference = 0.73, 95% CI 2-sided [0.00 to 1.46], Standard Error of Mean 0.371
Statistical Analysis 7: Comparison: Solifenacin 5 mg vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.011, ANCOVA; LS Mean Difference = 0.94, 95% CI 2-sided [0.22 to 1.66], Standard Error of Mean 0.368
Statistical Analysis 8: Comparison: Placebo vs Mirabegron 25 mg; Test type: Superiority or Other; p = 0.70, ANCOVA; LS Mean Difference = 0.17, 95% CI 2-sided [-0.67 to 1.01], Standard Error of Mean 0.428
Statistical Analysis 9: Comparison: Placebo vs Mirabegron 50 mg; Test type: Superiority or Other; p = 0.084, ANCOVA; LS Mean Difference = 0.73, 95% CI 2-sided [-0.10 to 1.56], Standard Error of Mean 0.423
Statistical Analysis 10: Comparison: Placebo vs Solifenacin 2.5 mg; Test type: Superiority or Other; p = 0.12, ANCOVA; LS Mean Difference = 0.66, 95% CI 2-sided [-0.18 to 1.49], Standard Error of Mean 0.425
Statistical Analysis 11: Comparison: Placebo vs Solifenacin 5 mg; Test type: Superiority or Other; p = 0.36, ANCOVA; LS Mean Difference = 0.34, 95% CI 2-sided [-0.39 to 1.06], Standard Error of Mean 0.369
Statistical Analysis 12: Comparison: Placebo vs Solifenacin 10 mg; Test type: Superiority or Other; p = 0.23, ANCOVA; LS Mean Difference = 0.52, 95% CI 2-sided [-0.32 to 1.36], Standard Error of Mean 0.428
Statistical Analysis 13: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.16, ANCOVA; LS Mean Difference = 0.52, 95% CI 2-sided [-0.21 to 1.25], Standard Error of Mean 0.371
Statistical Analysis 14: Comparison: Placebo vs Solifenacin 2.5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.032, ANCOVA; LS Mean Difference = 0.79, 95% CI 2-sided [0.07 to 1.52], Standard Error of Mean 0.371
Statistical Analysis 15: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.006, ANCOVA; LS Mean Difference = 1.03, 95% CI 2-sided [0.30 to 1.76], Standard Error of Mean 0.373
Statistical Analysis 16: Comparison: Placebo vs Solifenacin 5 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.031, ANCOVA; LS Mean Difference = 0.80, 95% CI 2-sided [0.07 to 1.52], Standard Error of Mean 0.369
Statistical Analysis 17: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 25 mg; Test type: Superiority or Other; p = 0.012, ANCOVA; LS Mean Difference = 1.07, 95% CI 2-sided [0.24 to 1.90], Standard Error of Mean 0.423
Statistical Analysis 18: Comparison: Placebo vs Solifenacin 10 mg + Mirabegron 50 mg; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = 1.28, 95% CI 2-sided [0.45 to 2.10], Standard Error of Mean 0.421

ADVERSE EVENTS:
Time Frame: Adverse events summarized for the Safety Analysis Set (SAF) were reported after the first dose of double-blind study drug and no more than 30 days after the last dose of double-blind study drug.
Description: The SAF included all patients randomized to a double-blind treatment who took at least 1 dose of study drug.One participant randomized to the Mirabegron 25 mg arm received treatment with Solifenacin 5 mg + Mirabegron 50 mg in error and is counted in that arm for safety analysis set analyses.
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 2.5 mg | Solifenacin 5 mg | Solifenacin 10 mg | Solifenacin 2.5 mg and Mirabegron 25 mg | Solifenacin 2.5 mg and Mirabegron 50 mg | Solifenacin 5 mg and Mirabegron 25 mg | Solifenacin 5 mg and Mirabegron 50 mg | Solifenacin 10 mg and Mirabegron 25 mg | Solifenacin 10 mg and Mirabegron 50 mg
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/77 | 2/78 | 1/79 | 0/156 | 1/78 | 3/149 | 2/149 | 2/144 | 2/153 | 1/81 | 1/81
Other Adverse Events (participants affected / at risk) | 16/81 | 16/77 | 21/78 | 19/79 | 48/156 | 33/78 | 36/149 | 34/149 | 40/144 | 39/153 | 30/81 | 35/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Mirabegron 25 mg (N=77) | Mirabegron 50 mg (N=78) | Solifenacin 2.5 mg (N=79) | Solifenacin 5 mg (N=156) | Solifenacin 10 mg (N=78) | Solifenacin 2.5 mg and Mirabegron 25 mg (N=149) | Solifenacin 2.5 mg and Mirabegron 50 mg (N=149) | Solifenacin 5 mg and Mirabegron 25 mg (N=144) | Solifenacin 5 mg and Mirabegron 50 mg (N=153) | Solifenacin 10 mg and Mirabegron 25 mg (N=81) | Solifenacin 10 mg and Mirabegron 50 mg (N=81)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fibrosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Mirabegron 25 mg (N=77) | Mirabegron 50 mg (N=78) | Solifenacin 2.5 mg (N=79) | Solifenacin 5 mg (N=156) | Solifenacin 10 mg (N=78) | Solifenacin 2.5 mg and Mirabegron 25 mg (N=149) | Solifenacin 2.5 mg and Mirabegron 50 mg (N=149) | Solifenacin 5 mg and Mirabegron 25 mg (N=144) | Solifenacin 5 mg and Mirabegron 50 mg (N=153) | Solifenacin 10 mg and Mirabegron 25 mg (N=81) | Solifenacin 10 mg and Mirabegron 50 mg (N=81)
Dry mouth (Gastrointestinal disorders) | 3 | 2 | 4 | 6 | 18 | 23 | 19 | 13 | 21 | 20 | 16 | 14
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 3 | 4 | 7 | 6 | 4 | 2 | 6 | 8
Nasopharyngitis (Infections and infestations) | 2 | 5 | 5 | 5 | 6 | 2 | 4 | 6 | 7 | 6 | 6 | 6
Escherichia urinary tract infection (Infections and infestations) | 2 | 1 | 2 | 1 | 6 | 5 | 3 | 2 | 3 | 4 | 3 | 1
Urinary tract infection (Infections and infestations) | 3 | 1 | 2 | 1 | 4 | 5 | 1 | 2 | 2 | 3 | 0 | 3
Hypertension (Vascular disorders) | 7 | 9 | 11 | 8 | 18 | 5 | 11 | 11 | 11 | 9 | 7 | 11

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 90 days prior to publication for review and comment.